CLINICAL TRIAL: NCT01307514
Title: Protocol for Evaluation of the Effects of Heating Massaging Vibrating or Application of Topical Agent on the Vicinity of the Insulin Delivery Site
Brief Title: Effects of Heating Massaging Vibrating Vicinity of the Insulin Delivery Site
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Raz, Hadassah Medical Organization
Other Study IDs: 0417-08-HMO
Record Dates: First submitted 2008-10-02; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2008-09

CONDITIONS: DIABETES
Keywords: DIABETES; PHARMACOKINETICS; PHARMACODYNAMICS; INSULIN
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The aim of this experiment is to test the pharmacodynamics and pharmacokinetics of insulin analogs and their dependence on external and physiological alterations. The investigators plan compare the pharmacodynamics of insulin analog delivery in regular conditions and in the presence of increased perfusion of the delivery site, achieved by way of local warming, movement and topical application of Capsaicin cream. The investigators will also test the effect of local heating and topical application of Capsaicin cream on the post prandial glucose levels following a bolus.

ELIGIBILITY:
Inclusion Criteria:

1. Participant age between 18- 65 years old
2. Type I or Type II diabetes
3. HbA1c 6-12%
4. Does not suffer from sever hypertension, kidney, liver or heart disease
5. Does not suffer from active Ischemic heart disease
6. Is willing to sign the consent form

Exclusion Criteria:

1. Participants age < 18 or > 65
2. Pregnancy
3. Breast feeding women
4. Un-controlled diabetes, HbA1c values > 12% range
5. Suffers from active Ischemic heart disease
6. Alcohol addiction
7. Is not prepared to signed the informed consent

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be patients with insulin dependent diabetes using standard insulin injections or continuous insulin infusion pumps.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel